CLINICAL TRIAL: NCT07011225
Title: Effects of Rehabilitation and Supplementation With Hydrolyzed Collagen vs. Whey Protein on the Cardiopulmonary, Renal, Muscular, and Immunohematological Response of COPD Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodolfo de Paula Vieira, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 7.040.417
Record Dates: First submitted 2025-03-11; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Collagen Supplementation; Whey Protein; Pulmonary Rehabilitation; COPD - Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary Inflammation; Pulmonary Rehabilitation; Dietary Supplementation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The volunteers will be randomly assigned to 4 groups, as follows: Control Group (GC; group only subjected to pre- and post-assessment; mild COPD n = 20; moderate COPD n = 20; severe COPD n = 20; very severe COPD n = 20), Whey Supplemented Group (GW; group supplemented with whey protein; mild COPD n = 20; moderate COPD n = 20; severe COPD n = 20; very severe COPD n = 20), Hydrolyzed Collagen Supplemented Group (GH; group supplemented with hydrolyzed collagen; mild COPD n = 20; moderate COPD n = 20; severe COPD n = 20; very severe COPD n = 20), Rehabilitation Group (GR; group subjected to rehabilitation; mild COPD n = 20; moderate COPD n = 20; severe COPD n = 20; very severe COPD n = 20). We clarify that the evaluations will be conducted before and after the rehabilitation period (nutritional supplementation).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Verisol Collagen 2.5 g/day (GCV) (Experimental): Supplementation with Verisol® collagen will be administered at a dose of 2.5 g/day, diluted in water or water-based juice (300-500 ml), and should be consumed daily for 7 days a week, over a period of 3 months.
  Interventions: Dietary Supplement: Verisol Collagen 2,5 g/day
- Peptech Collagen 2.5 g/day (GCP 2.5) (Experimental): Peptech® collagen will be administered at a dose of 2.5 g/day, diluted in water or water-based juice (300-500 ml), and should be consumed daily, 7 days a week, for 3 months.
  Interventions: Dietary Supplement: Peptech Collagen 2,5 g/day
- Peptech Collagen 10 g/day (GCP 10) (Experimental): Peptech® collagen supplementation at a dose of 10 g/day, diluted in water or water-based juice (300-500 ml), should be consumed daily, 7 days a week, for 3 months
  Interventions: Dietary Supplement: Peptech Collagen 10 g/day
- Group Control (Experimental): The control group will not receive any intervention during the first three months. After the evaluations, they will begin supplementation for an additional three months.
  Interventions: Diagnostic Test: Cardiorespiratory test
- Pulmonary rehabilitation with aerobic and resistance training. (Experimental)
  Interventions: Other: Pulmonary rehabilitation with aerobic and resistance training.

INTERVENTIONS:
Dietary Supplement: Verisol Collagen 2,5 g/day — Patients allocated to this group will consume Verisol Collagen 2,5 g/day for 90 days.
  Arms: Verisol Collagen 2.5 g/day (GCV)
Dietary Supplement: Peptech Collagen 2,5 g/day — Patients allocated to this group will consume Peptech Collagen 2,5 g/day for 90 days.
  Arms: Peptech Collagen 2.5 g/day (GCP 2.5)
Dietary Supplement: Peptech Collagen 10 g/day — Patients allocated to this group will consume Peptech Collagen 10 g/day for 90 days.
  Arms: Peptech Collagen 10 g/day (GCP 10)
Other: Pulmonary rehabilitation with aerobic and resistance training. — Patients enroled in this group will be submitted to Pulmonary rehabilitation with aerobic and resistance training.
  Arms: Pulmonary rehabilitation with aerobic and resistance training.
Diagnostic Test: Cardiorespiratory test — The patients allocated to this group will be submitted to initial and final evaluations only.
  Arms: Group Control

SUMMARY:
Chronic obstructive pulmonary disease (COPD) induces a severe loss of muscle strength and mass, in addition to reflecting significant pulmonary changes and causing cardiovascular, immunohematological, and renal alterations. In this regard, strategies capable of restoring or at least slowing the loss of muscle strength and mass are highly desirable. In this context, in addition to pulmonary rehabilitation with aerobic and strength exercises, supplementation with whey protein has been considered the gold standard for promoting muscle strength and mass gain in athletes. However, the potential effects of whey protein supplementation in patients with COPD remain unclear, which constitutes one of the objectives of the present study. A high percentage of elderly individuals present with lactose intolerance, milk protein allergies, or discomfort caused by components such as albumin, lactoferrin, casein, and alpha- and beta-globulin, making whey protein supplementation prohibitive for many elderly individuals, including those with COPD. Conversely, supplementation with collagen, particularly hydrolyzed collagen, offers a "pre-digested" protein option free from typical milk proteins. Additionally, the food industry has developed low molecular weight hydrolyzed collagen peptides, which may render such products hypoallergenic. To investigate these effects, 320 individuals aged 45 to 80 years with mild, moderate, severe, or very severe COPD (as defined by GOLD COPD 2025 criteria) will be recruited. Participants will be randomly assigned to four groups: Control Group (GC; subjected only to pre- and post-assessments; mild COPD n = 20; moderate COPD n = 20; severe COPD n = 20; very severe COPD n = 20), Whey Supplemented Group (GW; supplemented with whey protein; mild COPD n = 20; moderate COPD n = 20; severe COPD n = 20; very severe COPD n = 20), Hydrolyzed Collagen Supplemented Group (GH; supplemented with hydrolyzed collagen; mild COPD n = 20; moderate COPD n = 20; severe COPD n = 20; very severe COPD n = 20), and Rehabilitation Group (GR; subjected to rehabilitation; mild COPD n = 20; moderate COPD n = 20; severe COPD n = 20; very severe COPD n = 20). As outlined in the objectives and methodology of the project, the primary goals are to evaluate: (1) the effects of whey protein and (2) the effects of low molecular weight hydrolyzed collagen on pulmonary, cardiovascular, immunohematological, muscular, and renal parameters. The supplementation period will span three months, with evaluations conducted at baseline and after the supplementation period. Statistical analyses will be performed using the paired Student's t-test for intragroup comparisons and the unpaired Student's t-test for intergroup comparisons. A p-value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
As an inclusion criterion, patients with COPD must be included and must have been undergoing clinical-medication treatment for at least 90 days. As exclusion criteria, they should not have any type of autoimmune disease, must not be active smokers for at least 1 year, and in the case of ex-smokers, they must have quit smoking for at least 3 years, and must not have been engaging in any regular physical activity (˃1x/week) for at least 1 year.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentrations of Inflammatory and Regulatory Biomarkers | Baseline and after 3 months of intervention
  Plasma levels of IL-1β, IL-1ra, IL-6, IL-8, IL-10, IL-17, IL-23, IL-33, TNF-α, TGF-β, VEGF, and Klotho will be measured to evaluate the effect of supplementation with:
  10 g/day of whey protein isolate,
  2.5 g/day of Verisol® collagen,
  2.5 g/day of Peptech® collagen (low molecular weight peptides), and
  10 g/day of Peptech® collagen (low molecular weight peptides).
  Biomarkers will be quantified using enzyme-linked immunosorbent assay (ELISA) kits, following the manufacturer's instructions and international laboratory standards. Blood samples will be collected at two specific time points: baseline (prior to supplementation) and after three months of intervention.
  Data Aggregation: Mean and standard deviation of plasma concentrations for each biomarker within each group, with intra- and intergroup comparisons of pre- and post-intervention levels.

SECONDARY OUTCOMES:
Pulmonary Function Assessed by Spirometry | Baseline and after 3 months of intervention.
  Pulmonary function will be assessed using spirometry, following the parameters and guidelines established by the Sociedade Brasileira de Pneumologia e Tisiologia (SBPT). The following spirometric variables will be measured:
  Forced Vital Capacity (FVC),
  Forced Expiratory Volume in the first second (FEV1),
  FEV1/FVC ratio,
  Peak Expiratory Flow (PEF).
  Assessments will be performed at two specific time points: baseline (prior to supplementation) and after three months of intervention. Spirometry will be conducted by trained professionals using calibrated equipment, adhering to quality control standards recommended by the SBPT.
  Data Aggregation: Mean and standard deviation for each spirometric variable within each group, with intra- and intergroup comparisons of pre- and post-intervention values.
Cardiovascular Hemodynamics Assessed by PhysioFlow Impedance Cardiography | Baseline and after 3 months of intervention.
  Cardiovascular hemodynamics will be assessed non-invasively using PhysioFlow impedance cardiography. The following parameters will be measured: Stroke Volume and Stroke Volume Index, Cardiac Output and Cardiac Output Index, Early Diastolic Filling Ratio (Preload Index), and Systemic Vascular Resistance (Afterload). Assessments will be performed at two specific time points: baseline (prior to supplementation) and after three months of intervention. Measurements will be conducted by trained professionals using calibrated equipment, following the manufacturer's recommendations and quality control standards. Data will be aggregated as mean and standard deviation for each parameter within each group, with intra- and intergroup comparisons of pre- and post-intervention values.
  Data Aggregation: Mean and standard deviation for each cardiovascular parameter within each group, with intra- and intergroup comparisons of pre- and post-intervention values.

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelical University of Goiás, Anápolis, Goiás, Brazil